CLINICAL TRIAL: NCT06621602
Title: Quantification of Phosphorylated Alpha-synuclein in Cutaneous Biopsies as a Prospective Biomarker in Parkinson's Disease
Acronym: Syn-Q
Status: Active, not recruiting | Type: Observational
Sponsor: CND Life Sciences (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Other Study IDs: MJFF-025208
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: REM Behavior Disorder; Parkinson Disease
Keywords: PD; RBD
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue of the skin that is collected from three locations using a skin punch biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the levels of phosphorylated alpha-synuclein (P-SYN) in patients with Parkinson's disease and REM Behavior Disorder using a minimally invasive skin punch biopsy. It seeks to understand the natural progression of P-SYN deposition over time to explore the potential of P-SYN quantification as a biomarker for disease progression.

DETAILED DESCRIPTION:
This is a prospective, longitudinal study involving 75 Parkinson's disease patients and 25 patients with REM Behavior Disorder. Each participant will undergo a baseline evaluation followed by follow-ups every six months over an 18-month period. The evaluations will include clinical assessments, neurologic exams, and skin biopsies from three locations. Data will be collected on disease progression and the amount of P-SYN in cutaneous nerve fibers.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female 50 to 85 years of age
2. Clinical confirmed diagnosis of Parkinson's disease or REM Sleep Behavior

Exclusion Criteria:

1. Clinical evidence of severe vascular disease (history of ulceration, poor wound healing or vascular claudication)
2. History of allergic reaction to Lidocaine for local anesthesia needed for skin biopsies
3. Use of blood thinners (Plavix or Aspirin used separately is allowed)
4. Significantly impaired wound healing or history of scarring or keloid formation

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — sex at birth
Study Population: Subjects will be enrolled from 18 sites across the US from academic institutions and private clinics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Changes in phosphorylated alpha-synuclein and clinical assessments from Baseline at 18 months | 18 months
  The accuracy of the pathological test in detecting α-synuclein aggregation and deposition in skin punch biopsies.
  Measurement of the quantity of phosphorylated alpha-synuclein (P-SYN) in each biopsy to determine whether cutaneous biopsies can serve as a biomarker for changes in P-SYN deposition over time .
Changes in phosphorylated alpha-synuclein and clinical assessments from Baseline at 18 months | 18 months
  The precision of the pathological test in detecting α-synuclein aggregation and deposition in skin punch biopsies. Measurement of the quantity of phosphorylated alpha-synuclein (P-SYN) in each biopsy to determine whether cutaneous biopsies can serve as a biomarker for changes in P-SYN deposition over time .
  Time Frame: 18 months
Changes in phosphorylated alpha-synuclein and clinical assessments from Baseline at 18 months | 18 months
  The sensitivity of the pathological test in detecting α-synuclein aggregation and deposition in skin punch biopsies. Measurement of the quantity of phosphorylated alpha-synuclein (P-SYN) in each biopsy to determine whether cutaneous biopsies can serve as a biomarker for changes in P-SYN deposition over time . Time Frame: 18 months Time Frame: 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Todd Levine, Principal Investigator — CND Life Sciences
Locations (18):
- United States (18):
  - CND Life Sciences, Scottsdale, Arizona
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - Parkinson's Research Centers of America - Orange County, Aliso Viejo, California
  - Cedars Sinai, Los Angeles, California
  - Parkinson's Research Centers of America - Palo Alto, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - Aventura Neurologic Associates, LLC, Aventura, Florida
  - Parkinson's Disease and Movement Disorders Center - Boca Raton, Boca Raton, Florida
  - Atlanta NeuroScience Institute ANI, Atlanta, Georgia
  - Parkinson's Disease and Movement Disorders Center at KUMC, Kansas City, Kansas
  - Neurology Multidisciplinary Clinic at Norton Healthcare, Louisville, Kentucky
  - MedStar Montgomery Medical Center, Olney, Maryland
  - Boston Neuro Research Center, Boston, Massachusetts
  - Parkinson's Research Centers of America - Long Island, Commack, New York
  - University of Rochester, Rochester, New York
  - The Medical University of South Carolina, Charleston, South Carolina
  - Veracity Neuroscience LLC, Memphis, Tennessee
  - UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gibbons CH, Levine T, Adler C, Bellaire B, Wang N, Stohl J, Agarwal P, Aldridge GM, Barboi A, Evidente VGH, Galasko D, Geschwind MD, Gonzalez-Duarte A, Gil R, Gudesblatt M, Isaacson SH, Kaufmann H, Khemani P, Kumar R, Lamotte G, Liu AJ, McFarland NR, Miglis M, Reynolds A, Sahagian GA, Saint-Hillaire MH, Schwartzbard JB, Singer W, Soileau MJ, Vernino S, Yerstein O, Freeman R. Skin Biopsy Detection of Phosphorylated alpha-Synuclein in Patients With Synucleinopathies. JAMA. 2024 Apr 16;331(15):1298-1306. doi: 10.1001/jama.2024.0792. PMID 38506839